CLINICAL TRIAL: NCT06685250
Title: Randomized Controlled Trial Comparing Low (8 MmHg) Vs. Standard (14 MmHg) CO2 Insufflation Pressure on Postoperative Pain in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Postoperative Pain After a Laparoscopic Cholecystectomy
Acronym: CPOP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Charles Nicolle (Other)
Responsible Party: Principal Investigator, Dr Amine BEN SAFTA, surgical fellow in General Surgery, Hopital Charles Nicolle
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Chir-BS-2024-01
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pressure 8 mmHg (Experimental)
  Interventions: Procedure: Laparoscopic cholecystectomy
- Pressure 14 mmHg (Active Comparator)
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — Laparoscopic cholecystectomy

SUMMARY:
Randomized Controlled Trial to compare the effect of low (8 mmHg) versus Standard (14 mmHg) insufflation pressure of CO2 pneumoperitoneum on postoperative pain in patients undergoing laparoscopic cholecystectomy

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 or ASA 2
* uncomplicated symptomatic gallblader lithiasis scheduled for elective surgery
* no choledocholithiasis
* no associated surgical procedures
* no cerebrovasculare accident with neurological sequelae or other neurological disorders that affects sensation of pain
* no ascites
* no carcinomatosis

Exclusion Criteria:

* conversion to laparotomy
* need to keep an escat drain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2024-11-12 (Estimated); Primary Completion 2025-11-02 (Estimated); Study Completion 2025-12-02 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | Hour 6
  Visual Analog Scale (VAS) .from 0 to 10 0 no pain, 5 moderate pain, 10 worst possible pain

SECONDARY OUTCOMES:
postoperative pain | Hour 12
  Visual Analog Scale (VAS) 0 no pain, 10 worst possible pain
Postoperative pain | Hour 24
  Visual Analog Scale 0 no pain, 10 worst possible pain
vommiting (PONV score) | from 0 to 24 hours after surgery
  Postoperative Nausea and vomiting (PONV) score 0 no PONV , 1 moderate nausea, 2 moderate vomiting, 3 uncontrollable nausea and/or vomiting
morbidity | 30 days
postoperative length of stay | 30 days

REFERENCES:
- [Derived] Ben Safta A, Nasri S, Samaali I, Taher H, Trabelsi MM, Dziri C, Dougaz W, Nouira R. Randomized controlled trial comparing low pressure (8 mmHg) versus high pressure (14 mmHg) CO2 insufflation on postoperative pain in patients undergoing laparoscopic cholecystectomy: Protocol. PLoS One. 2025 Dec 18;20(12):e0339161. doi: 10.1371/journal.pone.0339161. eCollection 2025. PMID 41411326